CLINICAL TRIAL: NCT01606943
Title: The Study of The Chinese Registry of Acute Aortic Dissection and Clinical Study of Acute Aortic Dissection in Chinese Patients
Brief Title: Clinical Profiles and Outcomes of Acute Aortic Dissection in the Chinese Patients
Acronym: CPOAADCP
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Yang Li, MD, Principal Investigator, Xijing Hospital
Other Study IDs: XJ201202; CRAD2011 (Other Grant/Funding Number: 2011BAI11B00)
Record Dates: First submitted 2012-03-01; First posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Aorta Thoracic Ascending Dissection; Dissection of Descending Aorta
Keywords: Aortic dissection; Risk factor; Feature; Management; Outcome
MeSH Terms: conditions — Dissection, Thoracic Aorta; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clinical profiles and outcomes of patients with acute aortic dissection have not yet been evaluated in China. The aim of this study is to establish clinical registry of acute aortic dissection in China and to analyze clinical features, managements and outcomes of Chinese patients with acute aortic dissection.

DETAILED DESCRIPTION:
In 1996, the Internation Registry of Acute Aortic Dissection(IRAD) was established to improve clinical diagnosis and treatment of acute aortic dissection. However, most patients from the IRAD are Caucasian. These data were not sufficient to reflect clinical profiles and outcomes of Chinese patients with acute aortic dissection. In China, little is known about clinical features, managements and outcomes of acute aortic dissection involving a large number of patients. The investigators established clinical multicenter registry of acute aortic dissection. Between January 2009 and February 2012, about 2000 were enrolled in the Chinese registry of acute aortic dissection(CRAD) database. The aim of this study is to analyze clinical profiles and outcomes of Chinese patients with acute aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

* Stanford type A dissection
* Stanford type B dissection
* Retrograde Stanford Type B dissection
* Unclassified dissection with primary tear located in the aortic dissection

Exclusion Criteria:

* Aortic aneurysm
* Active infection or active vasculitides
* Myocardial infarction or Cerebral accident within 2 months
* Unwillingness to cooperate wiht study procedures or follow-up visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese population suffering acute aortic dissection
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dihua Yi, MD, Study Director — Xijing Hospital; Yang Li, MD, Principal Investigator — General Hospital of Beijing Military Area command of Chinese PLA; Wenxun Duan, MD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China